CLINICAL TRIAL: NCT06775249
Title: A Quick Mindfulness Training for an Isolated and Confined Environment (MINDFUL-ICE II)
Brief Title: A Quick Mindfulness Training for an Isolated and Confined Environment
Acronym: MINDFUL-ICE II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: ASI Agenzia Spaziale Italiana (Unknown); European Space Agency (ESA) (Unknown); Programma Nazionale di Ricerche in Antartide (PNRA) (Unknown); Institut Polaire Français Paul-Emile Victor (IPEV) (Unknown)
Responsible Party: Principal Investigator, Francesco Pagnini, Professor of Clinical Psychology, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CERPS_12-24
Record Dates: First submitted 2025-01-02; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Winter Crew At Concordia Station
Keywords: Isolated and Confined Environment; Mindfulness; Antarctica; Space Psychology

STUDY DESIGN:
Intervention Model Description: The study will use a quasi-experimental design with a quali-quantitative approach. Specifically, two winter-over crews will receive the mindfulness training, before and during the mission (experimental group). They will be assessed for stress, mindfulness, and psychosocial adaptation during the whole mission. Results will be compared with those collected during the MINDFUL-ICE study representing the control group. Moreover, participants will be monitored during the mission for their use of the intervention and will provide qualitative data about the usability and the efficacy of the mindfulness intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Training Program (Experimental): The intervention includes a three-week pre-departure online mindfulness course with bi-weekly booster sessions during the mission. Training focuses on stress reduction and fostering psychological flexibility, openness, and creativity.
  Interventions: Behavioral: ICE Mindfulness Program
- Historical data from MINDFUL-ICE I participants (No Intervention): The control group comprises data collected from participants in the MINDFUL-ICE I study (an observational cohort). These participants were winter-over crew members at Concordia Station, Antarctica, during earlier missions and did not receive any mindfulness-based intervention.

INTERVENTIONS:
Behavioral: ICE Mindfulness Program — The ICE Mindfulness Program is a tailored, self-paced intervention designed for crew members in isolated and confined environments. It includes a three-week pre-departure online course with videos, audio, and cognitive exercises promoting mindfulness, flexibility, and creativity, requiring 15-30 minutes daily. Delivered via email, it blends elements from Mindfulness-Based Stress Reduction and the Langerian approach. Participants receive new content daily, focusing on stress reduction and adaptation in extreme settings. Pre-departure, the PI leads a 1.5-hour interactive session with group meditation. During the mission, bi-weekly booster sessions are conducted by the ESA MD, supplemented by ongoing access to training materials. Exercises include meditations, mindful discussions, and cognitive tasks, with flexibility to fit participant schedules. The program will be available in Italian, French, and English.
  Arms: Mindfulness-Based Training Program

SUMMARY:
The MINDFUL-ICE II project explores the significance of mindfulness as a psychological trait crucial for extended missions in isolated and confined environments (ICEs). Previous data from the MINDFUL-ICE study with Concordia base crews validated a link between dispositional mindfulness and reduced stress. However, the efficacy of a mindfulness-based intervention in mitigating distress and fostering psychological adaptation within such environments remains untested. This project aims to assess a specific mindfulness training program's efficacy, feasibility, and usability for Concordia base crews over a two-year assignment. The pre-departure online mindfulness training, tailored for the pre-mission period, will feature minimal time commitments. Bi-weekly booster sessions during the mission, conducted by the ESA MD, will support the training. Using a quasi-experimental design, crews receiving this intervention will be compared with the first MINDFUL-ICE study's results. Stress, mindfulness, and psychological data will be tracked throughout the winter-over mission, aligning with the assessment approach of the initial study. Participants will report program usage, acquired knowledge, and engage in post-mission qualitative interviews. Both quantitative and qualitative findings will be crucial in gauging the intervention's effectiveness and usability for future long-duration and ICE space missions.

DETAILED DESCRIPTION:
Long-duration space missions introduce unique stressors, including isolation, confinement, communication delays, and environmental monotony, which can negatively affect mood, cognition, and performance. This study addresses the need for countermeasures by testing a mindfulness-based training program developed specifically for such environments. The intervention includes:

Pre-departure Training: A three-week, self-paced online course delivered via the Qualtrics platform, featuring videos, audio content, and exercises. Participants engage in daily activities averaging 15-30 minutes, focusing on mindfulness principles such as awareness, flexibility, and creativity.

Mission Phase: Bi-weekly booster sessions led by the ESA physician, supplemented by ongoing access to training materials. Content is tailored to address the challenges of ICE settings and can be accessed on-demand.

Assessment: Stress and mindfulness levels are measured at multiple time points (pre-departure, mid-mission, and post-mission). Additional qualitative feedback will explore participant experiences, training usability, and psychological adaptation.

The quasi-experimental design compares the outcomes of MINDFUL-ICE II participants with data from the previous observational MINDFUL-ICE study, which serves as a control group. This approach leverages matched cohorts to evaluate the program's efficacy in reducing stress and fostering adaptive psychological responses.

Data will be collected using validated psychometric tools, including the Perceived Stress Scale (PSS), Mindful Attention Awareness Scale (MAAS), and Langer Mindfulness Scale (LMS), alongside qualitative interviews and thematic analysis. Insights gained will contribute to the development of psychological interventions for future space exploration missions and other high-stress, isolated environments.

ELIGIBILITY:
Inclusion Criteria:

* Winter crew at the Concordia Station, in Antarctica

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Stress | Up to 12 months.
  Stress will be assessed using the Perceived Stress Scale, a validated 10-item self-report measure. Individual scores on the scale can range from 0 to 40 with higher scores indicating higher perceived.

SECONDARY OUTCOMES:
Mindful Attention | Up to 12 months.
  The Mindful Attention Awareness Scale: A 15-item self-report measure designed to assess a core characteristic of mindfulness, namely one's receptive awareness of and attention to what is taking place in the present. It has been validated in multiple languages, including Italian and French. The measure takes 5 minutes or less to complete. Based on a mean of all items, MAAS scores can range from 1 to 6. Higher scores indicate greater mindfulness.
Langerian Mindfulness | Up to 12 months.
  The Langer Mindfulness Scale: A 21-item questionnaire that assesses three domains describing mindful thinking: novelty seeking, engagement, flexibility, and novelty producing. It has been translated and validated in Italian, and the French validation is currently ongoing. The LMS can be completed in less than 5 minutes. The score ranges from to 21 to 147, with higher scores reflecting higher mindfulness.
Mindul Creativity | Up to 12 months (baseline and post-mission assessments).
  The Triangle Task assesses creative mindful thinking by asking participants to identify connections between abstract and concrete concepts (e.g., a "triangle" and related items). Scores reflect cognitive flexibility and openness. Scores range from 0 to 50, with higher scores reflecting higher mindful creativity.

OTHER OUTCOMES:
Program Engagement | Continuously during the mission, post-mission.
  The usage of the mindfulness exercises and other contents from the program will be continually monitored by (anonymously) tracking the access to the platform and with open-ended questions at every assessment time. These open-ended questions will ask how the participants used the mindfulness exercises and how they applied any mindset changes suggested by the training.
  An in-depth interview via video-call will be scheduled at the end of the mission to explore the perceived usefulness of the program and the qualitative impact of its contents. For example, participants will be asked if and how they applied contents and strategies from the program. They will also be asked how they dealt with possible crises, and whether they discussed some program contents with the fellow crewmembers.

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia Station, Antarctica, Antarctica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pagnini, F., Thoolen, S., Smith, N., Van Ombergen, A., Grosso, F., Langer, E., & Phillips, D. (2024). Mindfulness disposition as a protective factor against stress in Antarctica: A potential countermeasure for long-duration spaceflight?. Journal of Environmental Psychology, 94, 102254.